CLINICAL TRIAL: NCT02858986
Title: A Randomised Controlled Trial to Determine Whether a 3D Laparoscopic System Improves Surgeons' Performance During Laparoscopic Cholecystectomy When Compared to an Ultra-high Definition ('4K') Laparoscopic System
Brief Title: 3D Versus 4K Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Matt Dunstan, Surgical Research Registrar, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16SURN204848
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cholecystitis; Gallstones
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D laparoscopy (Experimental): Patients will undergo laparoscopic cholecystectomy using a 3D laparoscopic system
  Interventions: Procedure: 3D laparoscopy
- 4K laparoscopy (Experimental): Patients will undergo laparoscopic cholecystectomy using a 4K laparoscopic system
  Interventions: Procedure: 4K laparoscopy

INTERVENTIONS:
Procedure: 3D laparoscopy
  Arms: 3D laparoscopy
Procedure: 4K laparoscopy
  Arms: 4K laparoscopy

SUMMARY:
Introduction: Three-dimensional key-hole surgery ('laparoscopic') systems are proven to reduce the time required to complete tasks in laboratory settings. This benefit derives from the addition of binocular depth perception cues when compared to two-dimensional (2D) systems. This year a '4K' laparoscopic system has become commercially available, so-named as it provides a high resolution 2D image with four times the number of pixels of 2D full high definition. The improved visualisation is likely to provide additional non-binocular depth cues. It is currently unclear to what degree improving the resolution of 2D systems can compensate for binocular depth cues.

Aim: To determine whether the binocular vision provided by 3D laparoscopic systems provides benefits during laparoscopic cholecystectomy when compared to the monocular vision provided by high-resolution 4K systems.

Methods: A randomised controlled trial of 3D HD versus 4K laparoscopic systems will be performed, comparing the time to complete laparoscopic cholecystectomy, and error scores.

Impact: This study is a unique, first-of-its-kind investigation into two new surgical technologies, and is the first study to involve a 4K system. The uptake of three-dimensional systems has been curbed by financial cost and the limitations of early 3D technologies. This study aims to determine which system may be the safest, quickest and most cost- effective, in order to guide future investment and technological development towards either 3D or 2D systems. In addition, these systems may also aid in the learning curve of trainee surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Informed, written consent obtained after provision of information leaflets and face-to-face answering of any questions participants may have
2. Elective laparoscopic cholecystectomy
3. Medically fit for discharge as day case
4. Age 18 to 85 years

Exclusion Criteria:

1. Unable to obtain informed, written consent
2. Emergency cholecystectomy
3. Not medically fit for discharge as day case
4. Age <18 or >85 years
5. Conversion to open cholecystectomy
6. History of upper abdominal surgery
7. Recent/current involvement in another clinical trial
8. Common bile duct exploration at time of operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Time for completion of the key steps in laparoscopic cholecystectomy | Day of surgery

SECONDARY OUTCOMES:
Errors detected on video analysis of laparoscopic cholecystectomy as defined by a validated checklist | Day of surgery